CLINICAL TRIAL: NCT05743491
Title: A Feasibility Trial Comparing the Effectiveness of Yoga Versus Standard Care for Treating Fatigue in Hispanic Cancer Survivors
Brief Title: Yoga Versus Standard Care for Reducing Fatigue in Hispanic Cancer Survivors (YOCAS©®)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI moving to another institution
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Evelyn Arana, Research Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001111; UG1CA189961 (NIH); T32CA102618 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Fatigue; Cancer
MeSH Terms: conditions — Fatigue; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Experimental): Cancer survivors assigned to this condition continued with the standard follow-up care provided by their treating oncologists as appropriate for individual diagnoses. Participants in the control condition were offered the 4-week YOCAS©® program gratis after completing all study requirements.
  Interventions: Other: Standard Care
- YOCAS©® (Experimental): YOCAS©® is a standardized yoga program designed specifically for use by cancer patients and survivors. The YOCAS©® program is a low to moderate intensity mode of exercise that draws from two basic types of yoga: gentle Hatha and Restorative yoga. The program includes 18 specific physical postures (asanas) and mindfulness exercises focused on breathing (pranayama) and meditation (dhyana). The program is designed to be delivered by certified yoga instructors in community settings, two times a week for 75 minutes over four weeks.
  Interventions: Behavioral: YOCAS©®

INTERVENTIONS:
Other: Standard Care — Cancer survivors assigned to this condition continue with the standard follow-up care provided by their treating oncologists as appropriate for individual diagnoses. Participants in the control condition were offered the 4-week YOCAS©® program gratis after completing all study requirements.
  Other Names: Usual Care
  Arms: Standard Care
Behavioral: YOCAS©® — YOCAS©® is a standardized yoga program designed specifically for use by cancer patients and survivors. The YOCAS©® program is a low to moderate intensity mode of exercise that draws from two basic types of yoga: gentle Hatha and Restorative yoga. The program includes 18 specific physical postures (asanas) and mindfulness exercises focused on breathing (pranayama) and meditation (dhyana). The program is designed to be delivered by certified yoga instructors in community settings, two times a week for 75 minutes over four weeks.
  Arms: YOCAS©®

SUMMARY:
This is a phase II 2-arm randomized controlled trial comparing yoga (Yoga for Cancer Survivors, YOCAS©®) to standard care in reducing cancer-related fatigue in Hispanic cancer survivors. Survivors randomized to Arm 1 will receive Standard Care and Arm 2 will receive standard care plus a four-week YOCAS©® intervention where Hispanic survivors attend yoga sessions together. Investigators will acquire preliminary data on cancer-related fatigue, as well as, secondary data on other common side effects.

DETAILED DESCRIPTION:
Primary Aim:

To collect preliminary data comparing the effects of a YOCAS©® intervention to standard care on changes in cancer-related fatigue among Hispanic cancer survivors immediately post-intervention.

Secondary Aims:

A) To collect preliminary data comparing the effects of a YOCAS©® intervention to standard care on changes in quality of life and physical functioning.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm 1 = Participants undergo standard follow-up care provided by their treating oncologists as appropriate for individual diagnoses. Participants in the control condition are offered the 4-week YOCAS©® program gratis after completing all study requirements.

Arm 2 = Participants undergo the YOCAS©® intervention comprising 18 specific physical postures and mindfulness exercises focused on breathing and meditation and meet with the yoga instructor over 75 minutes 2 times a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have a confirmed diagnosis of solid tumor or hematologic malignancy
* Have completed all chemotherapy, surgery, and/or radiation therapy within the last 2 years
* Have a score ≥4 on a 0-10 fatigue screening scale
* Be at least 18 years of age
* Self-identify as Latino/a or Hispanic
* Be able to read and understand English or Spanish
* Be able to provide written informed consent
* Have the ability to attend 8 yoga sessions in-person

Exclusion Criteria:

* Have contraindications to yoga participation per their primary physician or oncologist
* Have practiced yoga within the 3 months prior to enrolling in the study
* Be planning to start yoga on their own during the time they are enrolled in the study
* Have distant metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Mean Change in Fatigue as Measured by the Multidimensional Fatigue Symptom Inventory-Short Form (MFSI-SF) Total Score Comparing YOCAS©® to Standard Care [Time Frame: Baseline up to post intervention (approximately 5 weeks) ] | Baseline to post intervention (approximately 5 weeks)
  The MFSI is a multidimensional 30-item fatigue scale developed specifically for documenting cancer-related fatigue. The total MFSI-SF score ranges from -24 to 96, with a higher score indicating a higher fatigue level.

SECONDARY OUTCOMES:
Mean Change in Quality of Life as measured by the Functional Assessment of Cancer Therapy-General (FACT-G) total score comparing YOCAS©® to Standard Care [Time Frame: Baseline up to post intervention (approximately 5 weeks) ] | Baseline to post intervention (approximately 5 weeks)
  The Functional Assessment of Cancer Therapy - General (FACT-G) is a 27-item questionnaire designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. The total FACT-G score ranges from 0-108 with a higher score indicating better quality of life.
Mean Change in Physical Functioning as Measured by the 30-second chair stand comparing YOCAS©® to Standard Care [Time Frame: Baseline up to post intervention (approximately 5 weeks) ] | Baseline to post intervention (approximately 5 weeks)
  The participant is instructed to sit in the middle of a chair, cross their arms over their chest, keep their feet flat on the floor, and repeatedly raise to stand up and sit back down on the chair for 30 seconds. The number of times patients come to a full standing position in 30 seconds is recorded.
Mean Change in Physical Functioning as Measured by the 30-second arm curl test comparing YOCAS©® to Standard Care [Time Frame: Baseline up to post intervention (approximately 5 weeks) ] | Baseline to post intervention (approximately 5 weeks)
  Participants are instructed to be seated on an upright chair and asked to repeatedly lift a 5 lb weight (for women) or an 8 lb weight (for men) for 30 seconds. The number of lifts in 30 seconds is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided